CLINICAL TRIAL: NCT03486210
Title: Pilot Suty of the Assessment of Food Preferences After Bariatric Surgery (BariaTaste Pilot)
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0694
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Food Preferences Variations Depending on Bariatric Surgery Status

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Phase 1 Group 1: Healthy volunteers
  Interventions: Behavioral: Food preference
- Phase 1 Group 2: Health professionals
  Interventions: Behavioral: Food preference
- Phase 2 Group 1: Control group : patients obese without surgery
  Interventions: Other: Psychological assesment
- Phase 2 Group 2: Patients who have underwent a sleeve gastrectomy
  Interventions: Other: Psychological assesment
- Phase 2 Group 3: Patients who have underwent a gastric bypass
  Interventions: Other: Psychological assesment

INTERVENTIONS:
Behavioral: Food preference — The study will take place in two phases. A first phase will consist in the validation of translations and the selection of images on 20 healthy volunteers and 20 health professionals specialized in nutrition. They will have to fill a form with images of food and evaluate to what extend they think the pictures represent what we can eat in France. This step will adapt the questionnaire to our country.
  Groups: Phase 1 Group 1; Phase 1 Group 2
Other: Psychological assesment — Phase performed with patients fasting for at least 2 hours before the different tests. The FLPQ will be compared between a group of patients suffering from unoperated obesity (OCt), a group of patients operated on a sleeve gastrectomy (OSl) and a group operated by a bypass (OBy) between 6 and 24 months post-surgery, randomized for the 6 combined tests (2 categories). The award can be made in 2 sessions of at least 3 of the 6 tests combined. Each test combines 2 of the 11 categories. The test will consist of 96 pairs of 16 food images presented on a computer screen in color. Participants will be invited to "choose the food they most want to eat", by pressing the corresponding computer button (choices saved by counting the frequency scores in E-prime).
  The level of hunger will be evaluated by an Analogical Visual Scale, ranging from 0 to 10.
  Patients should also complete 3 self-questionnaires used routinely (Binge Eating Scale, The Yale Food Addiction Scale, The UPPS-P short version).
  Groups: Phase 2 Group 1; Phase 2 Group 2; Phase 2 Group 3

SUMMARY:
More than 50,000 patients in France benefit from bariatric surgery every year. However, nutritional complications (protein malnutrition, hypoglycaemia) are common and primary or secondary weight failures (weight recovery) account for almost 20% of operated. Weight loss and the metabolic effects of surgery are not related only to a reduction in dietary intakes, but also to mechanisms independent of caloric reduction, such as eating behaviour after bariatric surgery (Gastric Bypass or sleeve gastrectomy). These choices are guided by perceived changes in the properties of the food, resulting in changes in tastes, palatability and more generally food preferences. Among available tools to evaluate dietary preferences we selected the Food Leeds Preference Questionnaire (FLPQ) to assess those modifications. During this test, photographs of food products classified according to predetermined characteristics are presented with different instructions and response design to estimate liking, wanted for food, implicitly or explicitly. Our main hypothesis is that the use of the Food Leeds Preference Questionnaire will highlight differences in dietary preferences according to the type of bariatric surgery performed.

We will be conducted a study observational study on three parallel groups: a control group composed of patients suffering from unoperated obesity, a group of patients operated for a sleeve gastrectomy and a group of patients operated for a gastric bypass. We will include 45 patients per group. The patients will have to pass the Leeds Food Preference Questionnaire (LFPQ). Our judgment criterion will be the degree of food preference assessed using the LFPQ. Participants will also be assessed on behavioural parameters with the Binge Eating Scale, the Yale Food Addiction Scale Version 2.0 and the Urgency, lack of Premeditation, lack of Perseverance and Sensation seeking Impulsive behavior scale (UPPS-P) short version.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, between 18 to 65 years old
* Patient with a BMI between 18.5 and 60 kg / m2: minimum 35 kg / m2 for the obesity group
* Patient undergoing initial assessment before bariatric surgery for the obesity group
* Patient being assessed for follow-up after bariatric surgery (after sleeve gastrectomy or gastric bypass)
* Patient agreeing to participate in the study.
* Patient affiliated to a Social Security scheme or beneficiary of such a scheme

Exclusion Criteria:

* Patient with other psychiatric comorbidities, including a bipolar mood disorder or eating disorder
* Patient with food eviction, whether medical or cultural
* Patient with ongoing psychotropic treatment (except anxiolytic treatment)
* Patient unable to give his agreement, not mastering the French language,
* Patient under authorship or curators

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will focus on a population of patients who are or have been obese and are being cared for at the Lyon Sud Hospital Center. Patients will either be undergoing initial assessment or being assessed for follow-up after bariatric surgery (after sleeve gastrectomy or gastric bypass).
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Degree of food preference | Day 1
  The degree of food preference will be measured using the Leeds Food Preference Questionnaire, that the investigator will have previously adapted in French for French population, in the form of counting frequency scores for each category of images.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain ICETA, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Lyon Sud, Pierre-Bénite, France